CLINICAL TRIAL: NCT06760611
Title: An Observational Cohort Analysis of Tissue Quality of Integra Dermal Matrix (Integra®)-Treated Burns and NovoSorb® Biodegradable Temporizing Matrix (BTM)-Treated Burns 12-36 Months Post Final Skin Graft Application
Brief Title: Tissue Quality of Integra vs. BTM Treated Burns
Status: Withdrawn | Type: Observational
Why Stopped: change in company prioritizations
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: T-IDRTTQ-001
Record Dates: First submitted 2024-11-19; First posted 2025-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Burn Injury; Burn Scar; Burn Wounds - Partial Thickness (2nd Degree); Skin Grafting
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — optional skin punch biopsy samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Integra Cohort: Patient with a burn treated with Integra® in conjunction with standard of care (SOC)* 12-36 months post final skin graft application. 25 unique cases will be enrolled into this group.
- BTM Cohort: Patient with a burn treated with BTM in conjunction with SOC* 12-36 months post- skin graft application. 25 unique cases will be enrolled into this group.
- Combination Cohort: Patient with a burn treated with Integra and BTM in different regions of the body in conjunction with SOC* 12-36 months post-skin graft application. Up to 10 unique cases can be enrolled into this group.

SUMMARY:
An observational analysis of Integra-treated burns and Novosorb Biodegradable Temporizing Matrix (BTM)-treated burns will be undertaken 12-36 months post final skin graft application by retrospectively analyzing the patient's electronic medical record, and prospectively using a non-invasive measures of tissue quality and patient-reported outcomes. Patients will be offered the option to consent for a tissue biopsy for pathological evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has reviewed the IRB-approved consent form, has been properly consented per the protocol and has documented their consent to participate in the study by signing the IRB-approved consent form.
2. Patient had a deep dermal or full-thickness burn that required skin grafting that was first treated with Integra* or BTM, and at least 70% 'take' followed by an autograft
3. Patient had final skin graft between 12-36 months prior enrollment in the study.
4. Burn must have been ≥10% total body surface area (TBSA) and ≤70% TBSA.
5. Patient is ≥ 21 years of age at the time of treatment.

Exclusion Criteria:

1. Patient had a radiation burn.
2. Patient was treated with Integra or BTM and closed via secondary intention.
3. Severe cognitive dysfunction or psychiatric disorders.
4. Immunocompromised patients.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to enroll a total of up to 60 subjects, with 25 unique patients in the Integra-treated burns cohort 25 unique patients in the BTM-treated burns cohort, and up to 10 unique patients in the combination arm
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Time from Integra or BTM treated burns to autograft procedure | 12-36 months post final skin graft application
  The primary evaluation of clinical use of Integra- and BTM-treated burns will be undertaken by assessing the time from device application to autograft procedure (time to graft).
Vancouver Scar Scale assessment of tissue quality | 12-36 months post final skin graft application
  Tissue quality will be assessed using the Vancouver Scar Scale (VSS) (to qualitatively measure scar quality) between an overall score of 0-13.
  A higher score on the VSS represents clinically worse scars.

SECONDARY OUTCOMES:
Length of Hospital Stays | 12-36 months post final skin graft application
  Length of hospital stay in days following treatment of burns with Integra or BTM
Number of complications | 12-36 months post final skin graft application
  Number complications (i.e. infection) in burns treated with Integra vs burns treated with BTM
Number of re-operations | 12-36 months post final skin graft application
  Number of re-operations in burns treated with Integra vs burns treated with BTM
Number of re-admissions | 12-36 months post final skin graft application
  Number of re-admissions in burns treated with Integra vs burns treated with BTM
Number of days in ICU | 12-36 months post final skin graft application
  Number of days in ICU of patients with burns treated with Integra vs burns treated with BTM
Percent of Integra or BTM 'take' | 12-36 months post final skin graft application
  Percent of Integra or BTM 'take' in burns treated with Integra vs burns treated with BTM
Time from admission to Integra or BTM application | 12-36 months post final skin graft application
  Time (number of days) from admission to Integra or BTM application to the burn
Autograft site details specifically associated with application of Integra or BTM on index injury | 12-36 months post final skin graft application
  Size, thickness, and mesh of autograft site specifically associated with application of Integra or BTM on index injury
Patient-Observer Scar Assessment Scale (POSAS) | 12-36 months post final skin graft application
  Qualitative evaluation of burns treated with Integra vs burns treated with BTM utilizing the POSAS.
  The POSAS total score ranges from 6 to 60. The lower score corresponds to a situation of normal skin and as scores increase, it corresponds to a situation different from normal skin/
Patient Survey Question regarding neuropathic pain | 12-36 months post final skin graft application
  Patient survey question regarding neuropathic pain in burns treated with Integra vs burns treated with BTM.
  Patient Survey Question: Do you experience neuropathic pain (numbness, pins and needles (tingling), or burning sensation) in your burn scar?
Tissue Pliability / Elasticity | 12-36 months post final skin graft application
  Use of a cutometer to measure tissue pliability / elasticity in burns treated with Integra vs burns treated with BTM.
Tissue Height | 12-36 months post final skin graft application
  Use of an ultrasound to measure tissue height in burns treated with Integra vs burns treated with BTM.
Tissue Density | 12-36 months post final skin graft application
  Use of an ultrasound to measure tissue density in burns treated with Integra vs burns treated with BTM.
Tissue Sensitivity | 12-36 months post final skin graft application
  Use of the Semmes-Weinstein Aesthesiometer to measure tissue sensitivity in burns treated with Integra vs burns treated with BTM.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Arnold, Study Director — Medical Affairs

IPD SHARING:
Plan to Share IPD: No